CLINICAL TRIAL: NCT03173508
Title: Effect of Acetazolamide on Right Ventricular Function at Rest in Patients With Chronic Obstructive Pulmonary Disease at Altitude. A Randomized, Placebo-controlled, Double-blind Parallel Trial
Brief Title: Effect of Acetazolamide on Right Ventricular Function at Rest in Patients With Respiratory Disease at Altitude
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2017-00137E
Record Dates: First submitted 2017-05-23; First posted 2017-06-01 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: right ventricular function; echocardiography; obstructive airway disease; emphysema; acetazolamide; altitude
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive; Emphysema | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACETAZOLAMIDE oral capsule (Active Comparator): Acetazolamide 375mg/day (capsule @125 mg: 1 in the morning, 2 in the evening), orally. Medication starts 24 hours before ascent to 3200m until the morning after the second night at 3200m
  Interventions: Drug: ACETAZOLAMIDE oral capsule
- PLACEBO oral capsule (Placebo Comparator): Placebo (capsules identically looking as acetazolamide capsules: 1 in the morning, 2 in the evening), orally. Medication starts 24 hours before ascent to 3200m until the morning after the second night at 3200m.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: ACETAZOLAMIDE oral capsule — Administration of 125mg acetazolamide in the morning, 250mg in the evening, starting 24 hours before departure to 3200m
  Arms: ACETAZOLAMIDE oral capsule
Drug: Placebo oral capsule — Administration of equally looking placebo capsules in the morning and evening, starting 24 hours before departure to 3200m
  Arms: PLACEBO oral capsule

SUMMARY:
This trial will evaluate the effect of acetazolamide (375 mg per day) vs. placebo on right ventricular function at acute altitude exposure in patients with COPD.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind parallel trial evaluating the effect of acetazolamide (375 mg per day) vs. placebo on right ventricular function at rest in lowlanders with chronic obstructive pulmonary disease travelling to altitude. Participants living in the Bishkek area, Kyrgyzstan (760m), will be transferred by car within 4h to the Tuja Ashu high altitude clinic (3200 m), and stay there for 2 days. Acetazolamide 375mg/day (or placebo) will be administered 24 hours before departure at 760 m and during the stay at altitude. Outcomes will be assessed during the stay at 3200 m.

Right ventricular function will be assessed by transthoracic echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, age 18-75 yrs.
* COPD diagnosed according to GOLD, FEV1 40-80% predicted, SpO2 ≥92% at 750 m.
* Born, raised and currently living at low altitude (<800m).
* Written informed consent.

Exclusion Criteria:

* COPD exacerbation, very severe COPD with hypoxemia at low altitude (FEV1/FVC <0.7, FEV1 <40% predicted, oxygen saturation on room air <92% at 750 m).
* Comorbidities such as uncontrolled cardiovascular disease, i.e., unstable systemic arterial hypertension, coronary artery disease; previous stroke; OSA; pneumothorax in the last 2 months.
* Internal, neurologic, rheumatologic or psychiatric disease including current heavy smoking (>20 cigarettes per day)
* Known renal failure or allergy to acetazolamide and other sulfonamides

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-02 (Actual)

PRIMARY OUTCOMES:
pulmonary artery pressure | Day 2 at 760m and 3200m
  Difference in altitude-induced change of pulmonary artery pressure (PAP) between acetazolamide and placebo group, measured by transthoracic echocardiography (tricuspid pressure gradient and pulmonary valve acceleration time)

SECONDARY OUTCOMES:
pulmonary artery pressure | Day 2 at 3200m
  Difference at altitude of pulmonary artery pressure (PAP) between acetazolamide and placebo group, measured by transthoracic echocardiography (tricuspid pressure gradient and pulmonary valve acceleration time)
cardiac output | Day 2 at 760m and 3200m
  Difference in altitude-induced change of cardiac output between acetazolamide and placebo group, measured by transthoracic echocardiography
cardiac output | Day 2 at 3200m
  Difference at altitude between acetazolamide and placebo group in cardiac output, measured by transthoracic echocardiography
right heart dimensions | Day 2 at 760m and 3200m
  Difference in altitude-induced change of right heart dimensions between acetazolamide and placebo group, measured by transthoracic echocardiography
right heart dimensions | Day 2 at 3200m
  Difference at altitude of right heart dimensions between acetazolamide and placebo group, measured by transthoracic echocardiography
right heart function | Day 2 at 760m and 3200m
  Difference in altitude-induced change of right heart function between acetazolamide and placebo group, measured by transthoracic echocardiography (TAPSE)
right heart function | Day 2 at 3200m
  Difference at altitude of right heart function between acetazolamide and placebo group, measured by transthoracic echocardiography (TAPSE)
stroke volume | Day 2 at 760m and 3200m
  Difference in altitude-induced change of stroke volume between acetazolamide and placebo group, measured by transthoracic echocardiography
stroke volume | Day 2 at 3200m
  Difference at altitude between acetazolamide and placebo group in stroke volume, measured by transthoracic echocardiography
volumes | Day 2 at 760m and 3200m
  Difference in altitude-induced change of volumes between acetazolamide and placebo group, measured by transthoracic echocardiography
volumes | Day 2 at 3200m
  Difference at altitude of volumes between acetazolamide and placebo group, measured by transthoracic echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ulrich, MD, Principal Investigator — University of Zurich; Talant M Sooronbaev, MD, Study Director — National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan
Locations (1):
- National Center for Cardiology and Internal Medicine, Bishkek, Kyrgyzstan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Preiss H, Mayer L, Furian M, Schneider SR, Muller J, Saxer S, Mademilov M, Titz A, Shehab A, Reimann L, Sooronbaev T, Tanner FC, Bloch KE, Ulrich S, Lichtblau M. Right ventricular strain impairment due to hypoxia in patients with COPD: a post hoc analysis of two randomised controlled trials. Open Heart. 2025 Jan 4;12(1):e002837. doi: 10.1136/openhrt-2024-002837. PMID 39756820